CLINICAL TRIAL: NCT00382057
Title: Effect of Increasing Testosterone Levels on Insulin Sensitivity in Men With the Metabolic Syndrome
Brief Title: Testosterone Effects on Men With the Metabolic Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5 K23 DK02858-1526; 5 K23 DK02858-02 6/15/05; 5K23DK002858-02 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-11

CONDITIONS: Metabolic Syndrome
Keywords: Testosterone; Insulin resistance; Insulin sensitivity; Metabolic disorders
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Metabolic Diseases | interventions — Testosterone; Anastrozole; Goserelin

INTERVENTIONS:
Drug: Testosterone
Drug: Anastrozole
Drug: Goserelin

SUMMARY:
The metabolic syndrome is a medical condition defined by high levels of cholesterol in the blood, high blood pressure, central obesity (gain in fat around the region of the stomach), and insulin resistance (body responds less well to insulin). This state of impaired insulin resistance can lead to type 2 diabetes mellitus, which is one of the most common metabolic disorders in the U.S. Numerous studies have shown an inverse relationship between insulin resistance and testosterone levels in men, however, causality has not been established. This protocol investigates the role of testosterone in modulating insulin sensitivity in insulin resistant states such as the metabolic syndrome. The hypothesis is that testosterone administration will improve insulin sensitivity.

DETAILED DESCRIPTION:
This protocol will address the impact of three months of testosterone (T) therapy on all components of the metabolic syndrome and the mechanism underlying changes in insulin sensitivity by analyzing changes in body composition, and detailed studies of fat metabolism and skeletal muscle. In addition, this protocol will address the role of estradiol (E2) in mediating the effect of testosterone on insulin sensitivity.

Seventy-two subjects will undergo a screening visit to assess eligibility after which a baseline evaluation will be performed. The baseline metabolic assessment will consist of an intravenous glucose tolerance test (IVGTT) to measure insulin sensitivity, MRI and DEXA scan to assess muscle and body fat distribution, VO2 max test and resting metabolic rate, and a muscle biopsy to look at how the muscle is affected by insulin and testosterone.

Subjects will then be randomized to one of three 12-week treatment arms, 1) Group 1 (Placebo); 2) Group 2 (Depot GnRH agonist (Zoladex) + T + placebo); or 3) Group 3 (Zoladex + T + aromatase inhibitor (anastrozole)). The rationale for this study design is as follows. Under normal physiological conditions, administration of T leads to a concomitant increase in E2 levels due to endogenous conversion by the aromatase enzyme system. Therefore, in order to dissect the relative roles of T and E2 on insulin sensitivity, one group of subjects will receive T in conjunction with the aromatase inhibitor, anastrozole.

At 13 weeks, the entire baseline evaluation including IVGTT, resting metabolic rate and VO2 max, body composition assessment by DEXA and MRI, and muscle biopsy will be repeated. Subjects will return for a follow up visit four weeks later to measure CBC, T and PSA levels, to ensure levels are within the normal range.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-75 yr
2. Diagnosis of the metabolic syndrome defined by the American Heart Association/National Heart, Lung, and Blood Institute guidelines as the presence of three or more of the following:

   * Waist circumference > 102 cm
   * Serum triglycerides > 150 mg/dL
   * HDL cholesterol < 40 mg/dL
   * Blood pressure > 130 mm Hg systolic or 85 mm Hg diastolic, or treatment with anti-hypertensives
   * Fasting serum glucose > 100 mg/dL
3. Plasma total testosterone level less than 300 ng/dL (1 SD below the mean for young healthy men)
4. Stable weight for previous three months (no weight change greater than or equal to +/-10 lbs)
5. Normal TSH, prolactin and prostate specific antigen (PSA) levels (<2.5 ng/mL)

Exclusion Criteria:

1. New diagnosis of type 2 diabetes as defined by the ADA criteria: fasting glucose greater than 126 mg/dL or random blood glucose greater than 200 mg/dL on two occasions, or on oral hypoglycemic agents
2. History of testicular disorders (i.e. cryptorchidism)
3. History of bleeding disorders (i.e. thrombocytopenia) or baseline hemoglobin levels less than 12g/dL
4. History of prostate cancer
5. History of sleep apnea (subjects will also be excluded if at their baseline assessment they admit to heavy snoring, restless sleep, and/or excessive daytime somnolence)
6. Symptoms of urinary outflow obstruction (i.e. benign prostatic hypertrophy)
7. Illicit drug use or heavy alcohol use (>4 drinks/day)
8. Allergic disorders
9. Current medications (must exclude individuals taking the following medications: Testosterone, Cimetidine, Spironolactone, Ketoconazole, Finasteride, DHEA, Androstenedione, Oral steroids, GnRH analogs)

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-05; Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity
muscle and body fat distribution
VO2 max
resting metabolic rate
muscle biopsy analysis

CONTACTS AND LOCATIONS:
Overall Officials: William F Crowley, MD, Study Director — Massachusetts General Hospital; Frances J Hayes, MD, Principal Investigator — Massachusetts General Hospital